CLINICAL TRIAL: NCT04976959
Title: High Fiber in Parkinson's Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Gian Dev Pal, MD, MS, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro2021000121
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Parkinson's patients (Experimental): Parkinson's patients who will receive a high fiber supplement
  Interventions: Drug: High Fiber supplement
- Control subjects (No Intervention): no supplement will be given

INTERVENTIONS:
Drug: High Fiber supplement — The supplement consists of a mixture of soluble fibers (from inulin and fibersol-2) and insoluble fibers (from oat bran, corn bran, wheat bran and sorghum bran) and it will be consumed as a drink.
  Arms: Parkinson's patients

SUMMARY:
The purpose of the research is to determine the effects of a high-fiber nutritional supplement (HFS) on the bacteria, viruses, and fungi that live in different regions of the body in those with Parkinson's disease (PD). We will compare the bacteria, viruses, and fungi of those with PD to those without PD (healthy controls). We will also examine the effects of transplanting stool from humans into laboratory mice with or without Parkinson-like pathology to understand how the microbiome influences the brains of animals. We can use this information to get a better understanding of how changing the microbiome might help humans.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patients who are untreated

Exclusion Criteria:

* Occupation expected to change the microbiome (e.g. sanitation worker)
* Treatment with medications that may induce parkinsonism (e.g. metoclopramide, typical or atypical antipsychotic agents)
* Treatment within 12 weeks with oral or intravenous antibiotics
* Known diagnosis of inflammatory bowel disease
* Symptomatic organic gastrointestinal (GI) disease (other than hemorrhoids and hiatal hernia) or abdominal surgeries for symptomatic gastrointestinal disease such as bowel resection, diverticular surgery, colostomy; subjects with a history of an appendectomy or gallbladder removal for non-cancerous disease more than 5 years prior to presentation are allowed.
* Symptomatic functional GI disease that significantly impairs intestinal motility such as scleroderma or use of GI motility drugs
* Acute illness requiring immediate hospitalization
* Pre-existent conditions as below:
* Liver disease (cirrhosis or persistently abnormal AST or ALT that are 2X> normal);
* Kidney disease (creatinine>2.0 mg/dL);
* Uncontrolled psychiatric illness;
* Clinically important lung disease or heart failure;
* HIV disease;
* Alcoholism, unreliable drinking history; or consumption of alcohol more than 3 times a week or binge drinking or drinking more than or equal to 3 drinks per occasion;
* Transplant recipients;
* Diabetes;
* BMI > 30
* Clinically significant dehydration or clinically detectable ascites or peripheral edema or cardiac failure
* Presence of short bowel syndrome or severe malnutrition with ideal body weight < or = 90%
* Use of immunosuppressive medications in 3 months prior to enrollment
* Anti-inflammatory medication use within 3 weeks of enrollment.
* Chronic use of diuretics

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
changes in microbiome composition | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gian Pal, MD, MS, Principal Investigator — Rutgers University
Locations (1):
- Rutgers-RWJ University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No